CLINICAL TRIAL: NCT00265174
Title: Serum DNA Analysis: Potential Application for Diagnosis and Prognosis in Brain Cancer.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: IRISL1-HMO-CTIL
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2005-12-14 (Estimated); Status verified 2005-11

CONDITIONS: Primary Brain Tumor
Keywords: SERUM DNA; LOH; METHYLATION; GLIOMA; MGMT
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
Numerous studies document the ability of tumors to shed DNA into the blood stream. Circulating DNA can thus be recovered for analyses, representing a surrogate tumor material to test for potential applications in disease diagnosis and prognosis.

Detection of genetic alternation is one of the most important tests for cancer patient since they offen correlated with the clinical course, prognosis and chemosensitivity of primary brain tumors. Currently in brain tumor patients these molecular aberrations can be analyzed only on tumor tissue that was obtained at surgery or biopsy.

Paucity of pathologic samples or poor fixation technique often make the tissue samples unassessable for molecular aberrations.

Therefore, the ability to extract tumor DNA from peripheral blood holds a great clinical significance. Still, the molecular aberration evaluated on serum DNA should be correlated and verified by comparison to standard evaluations performed on tumor samples. Our study aim is to evaluate the feasibility of using serum DNA for routine diagnosis of tumor molecular aberrations.

DETAILED DESCRIPTION:
Backround:

Genetic and epigenetic abrasions like loss of hetherozygosity and hypermethylation of gene promoters are common aberration in gliomas. Detection of these aberrations serves as diagnostic and prognostic tool. Examples: 1. oligodendrogliomas patients with combined 1p/19q LOH within the tumor respond better to chemotherapy and have better prognosis, whereas LOH on chromosome 10q is a marker for worse prognosis. 2. GBM patients with hypermethylation of the promoter of methyl-guanine-methyl-transferase (MGMT) in the tumor respond better to alkylating agent and have better prognosis.

As sample materials for diagnosis should be easily accessible by a minimally invasive procedure, there has been much interest in the potential use of nucleic acid markers in the blood of patients with cancer.

It was demonstrated that LOH as well as hypermethylation could be detected in the plasma/serum of patients with a variety of malignancies, suggesting that circulating tumor-associated DNA in the blood of patients can be a key determinant in predicting genetic and epigenetic abrasions in the tumor.

Objectives of the study:

Main objective: to find whether genetic abrasions in serum DNA represent the tumor DNA in patients with brain tumor.

Is tumor DNA can be detected in the serum of only high grade tumors or also in low grade tumor?

Methods:

Blood serum and tumor of patients are obtained anonymously, after the patient has signed a consent form, prior to surgery as part of the procedure for tissue collection for the brain tumor bank at Hadassah.

Part of the tumor is stained with hematoxylin-and-eosin and Histopathologic diagnosis is performed by a pathologist.

DNA is extracted from whole blood, serum and tumor of all patients with low grade or high grade gliomas.

In order to determine whether serum DNA represents the tumor DNA, LOH of 1p,19q,10q,17p,13q, 9p as well as methylation status of MGMT promoter will be tested in DNA samples from blood, serum and tumor.

ELIGIBILITY:
Inclusion Criteria:

LOW AND HIGH GRADE GLIOMAS

Exclusion Criteria:

NON GLIAL TUMORS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: TALI SIEGAL, MD, Principal Investigator — Hadassah Medical Organization; IRIS LAVON, PHD, Study Director — Hadassah Medical Organization
Locations (1):
- Hdassah Medical Organization, Jerusalem, Israel